CLINICAL TRIAL: NCT01460043
Title: Pilot Study of Homeopathy in Dysfunctional Uterine Bleeding Presenting as Menorrhagia
Brief Title: Trial of Homeopathy on Management of Menorrhagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMP-0032-HR
Record Dates: First submitted 2011-10-18; First posted 2011-10-26 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-10

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Homeopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Homeopathy (Experimental): Individualized symptom based therapy
  Interventions: Drug: Homeopathy

INTERVENTIONS:
Drug: Homeopathy — Each homeopathic medication was given as 1 g dose of homeopathic preparation in 30c potency. The dose is prepared as lactose globules on which the homeopathic preparation.
  Arms: Homeopathy
Drug: placebo — corresponding placebo was identical in appearance of homeopathic globule prepared in alcohol.
  Arms: placebo

SUMMARY:
The purpose of this study is to compare outcomes and quality-of-life issues in the treatment of menorrhagia, this randomized double blind controlled trial compared homeopathy and placebo. Clinical criteria were confirmed the diagnosis, and subjective assessment of the condition was performed during one pre-treatment and three treatment cycles. outcome measures were bleeding days, intensity. average pads used during menstrual cycle, abdominal & back pain, General health and overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35-49 years with regular heavy menstrual bleeding
* menstrual loss requiring more than 5 Pads/tampons per day
* menstrual cycle longer than 6 days

Exclusion Criteria:

* Organic causes of menorrhagia
* History of renal or hepatic impairment,
* Endocrine disorder including diabetes, thyroidism
* Thromboembolic disease,
* Inflammatory bowel disease,
* Peptic or intestinal ulceration, or coagulation or fibrinolytic disorders and --Malignancy.

Ages: 35 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
daily assessment of bleeding | change from baseline over 3 months
  bleeding days, intensity of bleeding, average pads used, back and abdominal pain associated.daily assessment during menses were completed by participants at baseline before randomization and at each menses for 3 month of intervention period.

SECONDARY OUTCOMES:
Health related quality of life | change from baseline over 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Principal Investigator — NMP Medical Research Institute